CLINICAL TRIAL: NCT00153322
Title: Shape Up Somerville: Eat Smart Play Hard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Tufts University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-OPHR-121519; R06 CCR 121519
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity; Community-based Participatory Research; School intervention; Parental Involvement
MeSH Terms: conditions — Pediatric Obesity

INTERVENTIONS:
Behavioral: Nurtition and Physical Activity Education

SUMMARY:
Community-based environmental approach to obesity prevention targeting first, second, and third grade students in Somerville, MA.

DETAILED DESCRIPTION:
This study will demonstrate using measures of effectiveness, the feasibility of partnering with the community to create, disseminate, implement and evaluate Shape Up Somerville: Eat Smart. Play Hard., a community-based environmental change intervention to prevent obesity in culturally diverse, high-risk, early elementary school children. Based on formative work with parents, children, teachers, school food service, school officials, and community members, a community-wide campaign will be developed with targeted environmental change strategies for early elementary school children within the before-, during-, and after-school environments reinforced by changes within the home and community to support behavioral action and maintenance. The intervention targeting children will bring the energy equation into balance by offering numerous physical activity options that total up to 125 kcals per day and by improving the composition of the food served and the dietary options, particularly snack foods, available throughout the day. This study will measure awareness and participation of the partners and residents within the community. In addition the temporal change in BMI z-score will be monitored internally in 700 Somerville children and externally in 1000 control children from 2 demographically-matched communities for one year and will be compared to the change in BMI z-score in children participating in Shape Up Somerville with children from control communities over the one-year intervention and for one year of follow up. If successful, Somerville will serve as the model community that paves the way for cost-effective nationwide environmental action to prevent obesity at the community level.

ELIGIBILITY:
Inclusion Criteria:

* Public school students in 1st, 2nd, and 3rd grade in Somerville, MA

Exclusion Criteria:

* none

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000
Dates: Start 2002-11; Study Completion 2005-06

PRIMARY OUTCOMES:
BMI at one year
Dietary Behavior at one year
Physical Activity Behavior at one year
Nutrition Policy and Infrastructure Outcomes

SECONDARY OUTCOMES:
Nutrition Policy and Infrastructure Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Christina D. Economos, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Friedman School of Nutrition, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Folta SC, Kuder JF, Goldberg JP, Hyatt RR, Must A, Naumova EN, Nelson ME, Economos CD. Changes in diet and physical activity resulting from the Shape Up Somerville community intervention. BMC Pediatr. 2013 Oct 4;13:157. doi: 10.1186/1471-2431-13-157. PMID 24093936